CLINICAL TRIAL: NCT04106492
Title: A Multicenter Phase 1/2a, Open-Label Study of SQ3370 in Patients With Advanced Solid Tumors
Brief Title: Phase 1/2a Study of SQ3370 in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Shasqi, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SQ3370-001; 2020-0185 (Other: MD Anderson Cancer Center)
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Results first posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Cancer
Keywords: Sarcoma; Cancer; Tumor; Soft Tissue Sarcoma; Solid Tumor; Doxorubicin; Intratumoral; Anthracycline; Phase 1; Ovarian Cancer; Precision Oncology; Precision Chemotherapy; Local Cancer Therapy; Targeted Cancer Therapy; Uterine Cancer; Head and Neck Cancer; Lung Cancer
MeSH Terms: conditions — Neoplasms; Sarcoma; Ovarian Neoplasms; Uterine Neoplasms; Head and Neck Neoplasms; Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase 1 dose escalation part of the study was done sequentially. The Phase 2 part of the study will be done in parallel between the four groups.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (15):
- Dose Escalation Cohort 1 (10 mL SQL70 and 8 mg/m^2 of SQP33) (Experimental): 10 mL of SQL70 injected intratumorally on Day 1 of each 21-day cycle into a single lesion with 8 mg/m^2 of SQP33 infused each day on Day 1 through Day 5 in subjects with locally advanced or metastatic solid tumors
  Interventions: Drug: SQ3370
- Dose Escalation Cohort 2 (10 mL SQL70 and 16 mg/m^2 of SQP33) (Experimental): 10 mL of SQL70 injected intratumorally on Day 1 of each 21-day cycle into a single lesion with 16 mg/m^2 of SQP33 infused each day on Day 1 through Day 5 in subjects with locally advanced or metastatic solid tumors.
  Interventions: Drug: SQ3370
- Dose Escalation Cohort 3 (10 mL SQL70 and 32 mg/m^2 of SQP33) (Experimental): 10 mL of SQL70 injected intratumorally on Day 1 of each 21-day cycle into a single lesion with 32 mg/m^2 of SQP33 infused each day on Day 1 through Day 5 in subjects with locally advanced or metastatic solid tumors.
  Interventions: Drug: SQ3370
- Dose Escalation Cohort 4 (10 mL SQL70 and 58 mg/m^2 of SQP33) (Experimental): 10 mL of SQL70 injected intratumorally on Day 1 of each 21-day cycle into a single lesion with 58 mg/m^2 of SQP33 infused each day on Day 1 through Day 5 in subjects with locally advanced or metastatic solid tumors.
  Interventions: Drug: SQ3370
- Dose Escalation Cohort 5 (10 mL SQL70 and 85 mg/m^2 of SQP33) (Experimental): 10 mL of SQL70 injected intratumorally on Day 1 of each 21-day cycle into a single lesion with 85 mg/m^2 of SQP33 infused each day on Day 1 through Day 5 in subjects with locally advanced or metastatic solid tumors
  Interventions: Drug: SQ3370
- Dose Escalation Cohort 6 (10 mL SQL70 and 125 mg/m^2 of SQP33) (Experimental): 10 mL of SQL70 injected intratumorally on Day 1 of each 21-day cycle into a single lesion with 125 mg/m^2 of SQP33 infused each day on Day 1 through Day 5 in subjects with locally advanced or metastatic solid tumors
  Interventions: Drug: SQ3370
- Dose Escalation Cohort 7 (10 mL SQL70 and 185 mg/m^2 of SQP33) (Experimental): 10 mL of SQL70 injected intratumorally on Day 1 of each 21-day cycle into a single lesion with 185 mg/m^2 of SQP33 infused each day on Day 1 through Day 5 in subjects with locally advanced or metastatic solid tumors
  Interventions: Drug: SQ3370
- Dose Escalation Cohort 8 (10 mL SQL70 and 250 mg/m^2 of SQP33) (Experimental): 10 mL of SQL70 injected intratumorally on Day 1 of each 21-day cycle into a single lesion with 250 mg/m^2 of SQP33 infused each day on Day 1 through Day 5 in subjects with locally advanced or metastatic solid tumors
  Interventions: Drug: SQ3370
- Dose Escalation Cohort 9 (10 mL SQL70 and 315 mg/m^2 of SQP33) (Experimental): 10 mL of SQL70 injected intratumorally on Day 1 of each 21-day cycle into a single lesion with 315 mg/m^2 of SQP33 infused each day on Day 1 through Day 5 in subjects with locally advanced or metastatic solid tumors
  Interventions: Drug: SQ3370
- Dose Escalation Cohort (20 mL SQL70 and 85 mg/m^2 of SQP33) (Experimental): 20 mL of SQL70 injected intratumorally on Day 1 of each 21-day cycle into a single lesion with 85 mg/m^2 of SQP33 infused each day on Day 1 through Day 5 in subjects with locally advanced or metastatic solid tumors
  Interventions: Drug: SQ3370
- Dose Escalation Cohort (20 mL SQL70 and 125 mg/m^2 of SQP33) (Experimental): 20 mL of SQL70 injected intratumorally on Day 1 of each 21-day cycle into a single lesion with 125 mg/m^2 of SQP33 infused each day on Day 1 through Day 5 in subjects with locally advanced or metastatic solid tumors
  Interventions: Drug: SQ3370
- Cohort A (10 mL SQL70 and 185 mg/m^2 of SQP33) (Experimental): 10 mL of SQL70 injected intratumorally on Day 1 of each 21-day cycle into a single lesion with 185 mg/m^2 of SQP33 infused each day on Day 1 through Day 5 in subjects with locally advanced or metastatic solid tumors
  Interventions: Drug: SQ3370
- P2a Group 1 (Extremity STS) (20 mL SQL70 and 250 mg/m^2/Day of SQP33) (Experimental): 20 mL of SQL70 injected intratumorally on Day 1 of each 21-day cycle into a single lesion with 250 mg/m^2 of SQP33 infused each day on Day 1 through Day 5 in subjects with soft tissue sarcomas of the extremity
  Interventions: Drug: SQ3370
- P2a Group 2 (10 mL SQL70 and 500 mg/m^2/ of SQP33 for 2 days and and 250 mg/m^2/ of SQP33 for 1 day) (Experimental): 10 mL of SQL70 injected intratumorally on Day 1 of each 21-day cycle into a single lesion with 500 mg/m^2 of SQP33 infused on Day 1 and 2 with 250 mg/m^2 of SQP33 infused on each Day 3 in subjects with locally advanced, unresectable or metastatic soft tissue sarcomas who are anthracycline naïve
  Interventions: Drug: SQ3370
- P2a Group 2 (10 mL SQL70 and 250 mg/m^2/day of SQP33 for five days) (Experimental): 10 mL of SQL70 injected intratumorally on Day with 250 mg/m^2 of SQP33 infused each day on Day 1 through Day 5 in subjects with locally advanced, unresectable or metastatic soft tissue sarcomas who are anthracycline naïve
  Interventions: Drug: SQ3370

INTERVENTIONS:
Drug: SQ3370 — SQ3370 consists of 2 components: SQL70, a protodrug-activating biopolymer, and SQP33, a protodrug of Doxorubicin

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and preliminary activity of SQ3370 in patients with advanced solid tumors.

ELIGIBILITY:
Phase 1: Inclusion Criteria:

1. Diagnosis of advanced soft tissue sarcoma or other solid tumors
2. Adequate hematologic, hepatic, renal, and coagulation function
3. ECOG performance status score 0-1
4. Tumor is the type where published clinical data would suggest that anthracyclines have cytotoxic activity
5. Injectable tumor present

Phase 1: Exclusion Criteria:

1. Prior exposure to 300 mg/m^2 of Dox HCl or DOXIL / CAELYX ® or 600 mg/m^2 of Epirubicin HCl
2. Congestive heart failure (CHF), severe myocardial insufficiency, or cardiac arrhythmia
3. Any of the following within 28 days prior to Cycle 1 Day 1:

   * Major surgery, as defined by the Investigator
   * Radiotherapy
   * Chemotherapy, immunotherapy and/or anticancer therapy (except for small molecule kinase inhibitors, which are 6 elimination half-lives)
4. Trastuzumab or trastuzumab emtansine dosed within 7 months prior to Cycle 1 Day 1.
5. Any transfusion within 14 days prior to Cycle 1 Day 1.
6. Pregnant or breast-feeding women.
7. Known active CNS metastases and/or carcinomatous meningitis or symptomatic brain metastasis. Participants with previously treated brain metastases may participate provided they are radiologically stable
8. History of allergic reactions attributed to Dox or other anthracyclines, NaHA, hyaluronic acid, or gram-positive bacterial proteins
9. History or evidence of clinically unstable/uncontrolled disorder, condition, or disease

Phase 2a Expansion Group 1 (Extremity STS): Inclusion

1. Patients with unresectable soft tissue sarcomas of the extremity AJCC Stage III OR select IV (=>5 cm injectable tumors) locally advanced and or metastatic, not amendable to primary surgical intervention according to the consensus of a multidisciplinary treatment team, determined prior to screening.
2. High grade STS, Grade 2/3, with an assessable/injectable lesion of at least diameter ≥5 cm by RECIST 1.1 criteria
3. No prior chemotherapy for STS, or radiation to affected limb

Phase 2a Expansion Group 1 (Extremity STS): Exclusion

1. Uncontrolled pain related to tumor
2. Open wounds or tissue necrosis related to tumor mass
3. Compartment syndrome or impending compartment syndrome

Phase 2a Expansion Group 2 (Unresectable STS): Inclusion

1. Locally advanced or metastatic, unresectable, soft-tissue sarcoma of intermediate or high grade with measurable disease.
2. Life expectancy >12 weeks (about 3 month)

Phase 2a Expansion Group 2 (Unresectable STS): Exclusion

1. Prior exposure to anthracyclines
2. Treatment naive extremity tumors

Phase 2a Expansion Group 3a (Head and Neck): Inclusion

1. Patients with histologically or cytologically confirmed squamous-cell carcinoma of the head and neck (HNSCC) who meet any of the following a) confirmed relapsed HNSCC or b) metastatic at initial presentation HNSCC
2. Patients who may have received two or less systemic regimens (therapies include chemotherapy and/or immunotherapy)

Phase 2a Expansion Group 3a (Head and Neck): Exclusion

1. Airway obstruction by tumor mass that requires clinical intervention
2. Prior treatment with anthracyclines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2023-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jim Williams, MD, Study Director — Shasqi, Inc.
Locations (10):
- United States (7):
  - City of Hope, Duarte, California
  - Stanford Cancer Center, Palo Alto, California
  - Sarcoma Oncology Center, Santa Monica, California
  - Washington University in St. Louis, St Louis, Missouri
  - Oregon Health & Science University, Portland, Oregon
  - MD Anderson Cancer Center, Houston, Texas
  - University of Washington, Seattle, Washington
- Australia (3):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Cancer Research Institute, Adelaide, South Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Srinivasan S, Yee NA, Aleckovic M, Zakharian M, Mahmoodi A, Wagner S, Nguyen TH, Chawla SP, Guminski AD, Mejia Oneto JM. Development of a First-in-Class Click Chemistry-Based Cancer Therapeutic, from Preclinical Evaluation to a First-in-Human Dose Escalation Clinical Trial. Clin Cancer Res. 2025 Sep 2;31(17):3662-3677. doi: 10.1158/1078-0432.CCR-24-2539. PMID 40522144
- [Derived] Srinivasan S, Yee NA, Zakharian M, Aleckovic M, Mahmoodi A, Nguyen TH, Mejia Oneto JM. SQ3370, the first clinical click chemistry-activated cancer therapeutic, shows safety in humans and translatability across species. bioRxiv [Preprint]. 2023 Mar 29:2023.03.28.534654. doi: 10.1101/2023.03.28.534654. PMID 37034617

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 2a Expansion Group 1 (Extremity STS) (20 mL SQL70 and 250 mg/m^2/Day of SQP33): 20 mL of SQL70 injected intratumorally on Day 1 of each 21-day cycle into a single lesion with 250 mg/m^2 of SQP33 infused each day on Day 1 through Day 5 in subjects with soft tissue sarcomas of the extremity
- P2a Grp 2 (10 mL SQL70 and 500 mg/m^2/ of SQP33 for 2 Days and and 250 mg/m^2/ of SQP33 for 1 Day): 10 mL of SQL70 injected intratumorally on Day 1 of each 21-day cycle into a single lesion with 500 mg/m^2 of SQP33 infused on Day 1 and 2 with 250 mg/m^2 of SQP33 infused on each Day 3 in subjects with locally advanced, unresectable or metastatic soft tissue sarcomas who are anthracycline naïve
- P2a Grp 2 (10 mL SQL70 and 250 mg/m^2/Day of SQP33 for Five Days): 10 mL of SQL70 injected intratumorally on Day with 250 mg/m^2 of SQP33 infused each day on Day 1 through Day 5 in subjects with locally advanced, unresectable or metastatic soft tissue sarcomas who are anthracycline naïve
Period: Overall Study
Arm/Group | Dose Escalation Cohort 1 (10 mL SQL70 and 8 mg/m^2 of SQP33) | Dose Escalation Cohort 2 (10 mL SQL70 and 16 mg/m^2 of SQP33) | Dose Escalation Cohort 3 (10 mL SQL70 and 32 mg/m^2 of SQP33) | Dose Escalation Cohort 4 (10 mL SQL70 and 58 mg/m^2 of SQP33) | Dose Escalation Cohort 5 (10 mL SQL70 and 85 mg/m^2 of SQP33) | Dose Escalation Cohort 6 (10 mL SQL70 and 125 mg/m^2 of SQP33) | Dose Escalation Cohort 7 (10 mL SQL70 and 185 mg/m^2 of SQP33) | Dose Escalation Cohort 8 (10 mL SQL70 and 250 mg/m^2 of SQP33) | Dose Escalation Cohort 9 (10 mL SQL70 and 315 mg/m^2 of SQP33) | Dose Escalation Cohort (20 mL SQL70 and 85 mg/m^2 of SQP33) | Dose Escalation Cohort (20 mL SQL70 and 125 mg/m^2 of SQP33) | Cohort A (10 mL SQL70 and 185 mg/m^2 of SQP33) | Phase 2a Expansion Group 1 (Extremity STS) (20 mL SQL70 and 250 mg/m^2/Day of SQP33) | P2a Grp 2 (10 mL SQL70 and 500 mg/m^2/ of SQP33 for 2 Days and and 250 mg/m^2/ of SQP33 for 1 Day) | P2a Grp 2 (10 mL SQL70 and 250 mg/m^2/Day of SQP33 for Five Days)
Started | 1 | 1 | 1 | 3 | 3 | 4 | 4 | 7 | 6 | 5 | 3 | 1 | 2 | 6 | 6
Completed | 1 | 1 | 1 | 3 | 3 | 4 | 4 | 7 | 6 | 5 | 3 | 1 | 2 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Cohort 1 (10 mL SQL70 and 8 mg/m^2 of SQP33) | Dose Escalation Cohort 2 (10 mL SQL70 and 16 mg/m^2 of SQP33) | Dose Escalation Cohort 3 (10 mL SQL70 and 32 mg/m^2 of SQP33) | Dose Escalation Cohort 4 (10 mL SQL70 and 58 mg/m^2 of SQP33) | Dose Escalation Cohort 5 (10 mL SQL70 and 85 mg/m^2 of SQP33) | Dose Escalation Cohort 6 (10 mL SQL70 and 125 mg/m^2 of SQP33) | Dose Escalation Cohort 7 (10 mL SQL70 and 185 mg/m^2 of SQP33) | Dose Escalation Cohort 8 (10 mL SQL70 and 250 mg/m^2 of SQP33) | Dose Escalation Cohort 9 (10 mL SQL70 and 315 mg/m^2 of SQP33) | Dose Escalation Cohort (20 mL SQL70 and 85 mg/m^2 of SQP33) | Dose Escalation Cohort (20 mL SQL70 and 125 mg/m^2 of SQP33) | Cohort A (10 mL SQL70 and 185 mg/m^2 of SQP33) | Phase 2a Expansion Group 1 (Extremity STS) (20 mL SQL70 and 250 mg/m^2/Day of SQP33) | P2a Grp 2 (10 mL SQL70 and 500 mg/m^2/ of SQP33 for 2 Days and and 250 mg/m^2/ of SQP33 for 1 Day) | P2a Grp 2 (10 mL SQL70 and 250 mg/m^2/Day of SQP33 for Five Days) | Total
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 3 | 4 | 4 | 7 | 6 | 5 | 3 | 1 | 2 | 6 | 6 | 53
Age, Continuous [Median (Full Range); unit: years] | 66 [66 to 66] | 70 [70 to 70] | 47 [47 to 47] | 65 [45 to 77] | 68 [45 to 79] | 44.5 [26 to 58] | 63.5 [54 to 73] | 65 [35 to 92] | 62 [31 to 78] | 63 [36 to 84] | 53 [23 to 76] | 84 [84 to 84] | 45 [32 to 58] | 64 [47 to 89] | 57 [45 to 69] | 58 [23 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 1 | 1 | 3 | 3 | 4 | 4 | 4 | 0 | 1 | 1 | 2 | 2 | 27
  Male | 1 | 1 | 0 | 2 | 2 | 1 | 1 | 3 | 2 | 1 | 3 | 0 | 1 | 4 | 4 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 2 | 0 | 0 | 2 | 0 | 1 | 10
  Not Hispanic or Latino | 1 | 1 | 1 | 3 | 3 | 3 | 3 | 4 | 6 | 3 | 3 | 1 | 0 | 6 | 5 | 43
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 1 | 1 | 1 | 3 | 1 | 4 | 4 | 6 | 5 | 4 | 3 | 1 | 2 | 4 | 5 | 45
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 1 | 0 | 1 | 1 | 1 | 2 | 3 | 6 | 5 | 5 | 3 | 1 | 2 | 6 | 5 | 42
  Australia | 0 | 1 | 0 | 2 | 2 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 11
Prior exposure to anthracyclines [Count of Participants; unit: Participants] | 0 | 1 | 0 | 2 | 2 | 1 | 2 | 3 | 1 | 4 | 3 | 0 | 0 | 0 | 0 | 19

OUTCOME MEASURES:

1. Primary Outcome: Phase 1 Cohorts
Description: To determine the Recommended Phase 2 Dose of SQ3370
Time Frame: From start of treatment to approximately 12 weeks
Population: Dose escalation participants
Measure: Number; unit: mg/m2 per cycle
Groups:
- Dose Escalation Cohort (10 mL SQL70): Participants will receive 10 mL of SQL70 biopolymer injected intratumorally on Day 1 of each 21-day cycle into a single lesion and then receive escalating doses of SQP33 protodrug administered IV from Day 1 through Day 5 (5 doses) of each 21-day cycle.
  SQ3370: SQ3370 consists of 2 components: SQL70, a protodrug-activating biopolymer, and SQP33, a protodrug of Doxorubicin
- Dose Escalation Cohort (20 mL SQL70): Participants will receive 20 mL of SQL70 biopolymer injected intratumorally on Day 1 of each 21-day cycle into a single lesion and then receive escalating doses of SQP33 protodrug administered IV from Day 1 through Day 5 (5 doses) of each 21-day cycle.
  SQ3370: SQ3370 consists of 2 components: SQL70, a protodrug-activating biopolymer, and SQP33, a protodrug of Doxorubicin
Arm/Group | Dose Escalation Cohort (10 mL SQL70) | Dose Escalation Cohort (20 mL SQL70)
Number analyzed (Participants) | 30 | 8
mg/m2 per cycle | 1250 | 1250

2. Secondary Outcome: Phase 2a: Objective Response Rate (ORR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 1 year
Measure: Number; unit: participants with an objective response
Groups:
- Cohort A (10 mL SQL70 and 185 mg/m2/Day of SQP33): Participants will receive SQL70 biopolymer injected intratumorally on Day 1 of each 21-day cycle into a single lesion as determined in Dose Escalation. Then will receive a lower dose than RP2D of SQP33 protodrug administered IV from Day 1 through Day 5 (5 doses) of each 21-day cycle.
  SQ3370: SQ3370 consists of 2 components: SQL70, a protodrug-activating biopolymer, and SQP33, a protodrug of Doxorubicin
- Phase 2a Expansion Group 1 (Extremity STS) (10 mL SQL70 and 250 mg/m2/Day of SQP33): Participants with soft tissue sarcomas of the extremity AJCC Stage III OR IV (>5 cm injectable tumors locally advanced and or metastatic, not amendable to primary surgical intervention and who are anthracycline naïve.
  SQ3370: SQ3370 consists of 2 components: SQL70, a protodrug-activating biopolymer, and SQP33, a protodrug of Doxorubicin
Arm/Group | Cohort A (10 mL SQL70 and 185 mg/m2/Day of SQP33) | Phase 2a Expansion Group 1 (Extremity STS) (10 mL SQL70 and 250 mg/m2/Day of SQP33) | P2a Grp 2 (10 mL SQL70 and 500 mg/m^2/ of SQP33 for 2 Days and and 250 mg/m^2/ of SQP33 for 1 Day) | P2a Grp 2 (10 mL SQL70 and 250 mg/m^2/Day of SQP33 for Five Days)
Number analyzed (Participants) | 1 | 2 | 6 | 6
participants with an objective response | 0 | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Dose Escalation Cohort 1 (10 mL SQL70 and 8 mg/m^2 of SQP33) | Dose Escalation Cohort 2 (10 mL SQL70 and 16 mg/m^2 of SQP33) | Dose Escalation Cohort 3 (10 mL SQL70 and 32 mg/m^2 of SQP33) | Dose Escalation Cohort 4 (10 mL SQL70 and 58 mg/m^2 of SQP33) | Dose Escalation Cohort 5 (10 mL SQL70 and 85 mg/m^2 of SQP33) | Dose Escalation Cohort 6 (10 mL SQL70 and 125 mg/m^2 of SQP33) | Dose Escalation Cohort 7 (10 mL SQL70 and 185 mg/m^2 of SQP33) | Dose Escalation Cohort 8 (10 mL SQL70 and 250 mg/m^2 of SQP33) | Dose Escalation Cohort 9 (10 mL SQL70 and 315 mg/m^2 of SQP33) | Dose Escalation Cohort (20 mL SQL70 and 85 mg/m^2 of SQP33) | Dose Escalation Cohort (20 mL SQL70 and 125 mg/m^2 of SQP33) | Cohort A (10 mL SQL70 and 185 mg/m^2 of SQP33) | Phase 2a Expansion Group 1 (Extremity STS) (20 mL SQL70 and 250 mg/m^2/Day of SQP33) | P2a Grp 2 (10 mL SQL70 and 500 mg/m^2/ of SQP33 for 2 Days and and 250 mg/m^2/ of SQP33 for 1 Day) | P2a Grp 2 (10 mL SQL70 and 250 mg/m^2/Day of SQP33 for Five Days)
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/1 | 0/1 | 0/3 | 0/3 | 0/4 | 0/4 | 0/7 | 0/6 | 0/5 | 0/3 | 0/1 | 0/2 | 1/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/1 | 1/1 | 2/3 | 2/3 | 0/4 | 2/4 | 2/7 | 0/6 | 1/5 | 1/3 | 0/1 | 0/2 | 2/6 | 1/6
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 3/3 | 3/3 | 4/4 | 4/4 | 7/7 | 6/6 | 5/5 | 3/3 | 1/1 | 2/2 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation Cohort 1 (10 mL SQL70 and 8 mg/m^2 of SQP33) (N=1) | Dose Escalation Cohort 2 (10 mL SQL70 and 16 mg/m^2 of SQP33) (N=1) | Dose Escalation Cohort 3 (10 mL SQL70 and 32 mg/m^2 of SQP33) (N=1) | Dose Escalation Cohort 4 (10 mL SQL70 and 58 mg/m^2 of SQP33) (N=3) | Dose Escalation Cohort 5 (10 mL SQL70 and 85 mg/m^2 of SQP33) (N=3) | Dose Escalation Cohort 6 (10 mL SQL70 and 125 mg/m^2 of SQP33) (N=4) | Dose Escalation Cohort 7 (10 mL SQL70 and 185 mg/m^2 of SQP33) (N=4) | Dose Escalation Cohort 8 (10 mL SQL70 and 250 mg/m^2 of SQP33) (N=7) | Dose Escalation Cohort 9 (10 mL SQL70 and 315 mg/m^2 of SQP33) (N=6) | Dose Escalation Cohort (20 mL SQL70 and 85 mg/m^2 of SQP33) (N=5) | Dose Escalation Cohort (20 mL SQL70 and 125 mg/m^2 of SQP33) (N=3) | Cohort A (10 mL SQL70 and 185 mg/m^2 of SQP33) (N=1) | Phase 2a Expansion Group 1 (Extremity STS) (20 mL SQL70 and 250 mg/m^2/Day of SQP33) (N=2) | P2a Grp 2 (10 mL SQL70 and 500 mg/m^2/ of SQP33 for 2 Days and and 250 mg/m^2/ of SQP33 for 1 Day) (N=6) | P2a Grp 2 (10 mL SQL70 and 250 mg/m^2/Day of SQP33 for Five Days) (N=6)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhagic transformation stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin T increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prohormone brain natriuretic peptide increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation Cohort 1 (10 mL SQL70 and 8 mg/m^2 of SQP33) (N=1) | Dose Escalation Cohort 2 (10 mL SQL70 and 16 mg/m^2 of SQP33) (N=1) | Dose Escalation Cohort 3 (10 mL SQL70 and 32 mg/m^2 of SQP33) (N=1) | Dose Escalation Cohort 4 (10 mL SQL70 and 58 mg/m^2 of SQP33) (N=3) | Dose Escalation Cohort 5 (10 mL SQL70 and 85 mg/m^2 of SQP33) (N=3) | Dose Escalation Cohort 6 (10 mL SQL70 and 125 mg/m^2 of SQP33) (N=4) | Dose Escalation Cohort 7 (10 mL SQL70 and 185 mg/m^2 of SQP33) (N=4) | Dose Escalation Cohort 8 (10 mL SQL70 and 250 mg/m^2 of SQP33) (N=7) | Dose Escalation Cohort 9 (10 mL SQL70 and 315 mg/m^2 of SQP33) (N=6) | Dose Escalation Cohort (20 mL SQL70 and 85 mg/m^2 of SQP33) (N=5) | Dose Escalation Cohort (20 mL SQL70 and 125 mg/m^2 of SQP33) (N=3) | Cohort A (10 mL SQL70 and 185 mg/m^2 of SQP33) (N=1) | Phase 2a Expansion Group 1 (Extremity STS) (20 mL SQL70 and 250 mg/m^2/Day of SQP33) (N=2) | P2a Grp 2 (10 mL SQL70 and 500 mg/m^2/ of SQP33 for 2 Days and and 250 mg/m^2/ of SQP33 for 1 Day) (N=6) | P2a Grp 2 (10 mL SQL70 and 250 mg/m^2/Day of SQP33 for Five Days) (N=6)
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 2 | 3 | 1 | 4 | 3 | 2 | 2 | 0 | 1 | 5 | 6
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 3 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 0 | 0 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colonic Fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Lip Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 3 | 1 | 1 | 1 | 3 | 4 | 1 | 1 | 0 | 2 | 2 | 4
Pyrexia (General disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Catheter Site Erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Face Oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
General Physical Health Deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Impaired Healing (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection Site Bruising (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection Site Erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Injection Site Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Medical Device Site Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 1 | 4 | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 2 | 0 | 0 | 1 | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bicytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 3 | 2 | 2 | 0 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Oral Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Candida Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Device Related Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Lymphangitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Medical Device Site Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular Access Site Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal Mycotic Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes Zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breast Pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic Pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blindness Transient (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry Eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Cardiac Failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bladder Spasm (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urge Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral Disc Displacement (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 0 | 0 | 0 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash Macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental Status Changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
Neuropathy Peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhagic Transformation Stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic Venous Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot Flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral Arterial Occlusive Disease (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular Access Site Erythema (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular Access Site Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb Injury (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Post Procedural Discharge (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vascular Access Site Pain (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-11-17): https://cdn.clinicaltrials.gov/large-docs/92/NCT04106492/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-19): https://cdn.clinicaltrials.gov/large-docs/92/NCT04106492/SAP_001.pdf